CLINICAL TRIAL: NCT01005563
Title: Effects of Dietary Protein Intake From Beef/Pork and Soy/Legumes on Appetite, Mood, and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0905008129; 0905008129 (Other: IRB Purdue University)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Appetite; Mood; Weight Loss
MeSH Terms: conditions — Weight Loss

ARMS (2):
- Arm 1: Beef/Pork (Experimental): Participants consuming diet with beef/pork as predominate sources of protein
  Interventions: Other: Beef/Pork
- Arm 2: Soy/Legumes (Experimental): Participants consuming diet with soy/legumes as predominate sources of protein
  Interventions: Other: Soy/Legumes

INTERVENTIONS:
Other: Beef/Pork — Participants consuming diet containing 10, 20 or 30% dietary protein with beef/pork as the predominate sources of protein
  Arms: Arm 1: Beef/Pork
Other: Soy/Legumes — Participants consuming diet containing 10, 20, or 30% dietary protein with soy/legumes as the predominate sources of protein.
  Arms: Arm 2: Soy/Legumes

SUMMARY:
The primary aims of this study are to assess the effects of habitual dietary protein intakes across the acceptable macronutrient distribution range with lean beef/pork or soy/legumes as the predominate sources of protein on indices of daily appetite and mood, and on postprandial appetite, mood, energy expenditure, and glycemic responses during energy-restricted weight loss in overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 21 years and older
* Body mass index between 27.0-36.9 kg/m2
* Non-smoking (within the last 6 months)
* Weight stable (< 3 kg (~7 lbs) weight gain or loss within last 3 months)
* Energy need for weight maintenance 1950-2750 kcal/day
* Not dietary restrained
* Menstruating women not pregnant or lactating
* Constant habitual activity patterns (within last 3 months)
* No Acute Illness (or have chronic diseases known to influence protein or energy metabolism)
* Non-diabetic
* Clinically normal blood profiles (within 10% of clinical normalcy)
* Non-hypertensive
* Not taking medications known to influence appetite or metabolism
* Willingness to eat study foods
* Able to travel to testing facility

Exclusion Criteria:

* Age: <21 years
* Body mass index: outside of the 27.0-36.9 kg/m2 range
* Smoker (currently or within the last 6 months)
* Gained or lost > 3.0 kg (7 lbs) within the last 3 months
* Energy need for weight maintenance < 1950 or > 2750 kcal/day
* Dietary restrained (≥ 14 on Three Factor Eating Questionnaire)
* Pregnant, lactating, or non-menstruating women
* Clinically diagnosed as a diabetic, or with liver or kidney disease/dysfunction, or osteoporosis
* Clinically abnormal blood profiles as identified by our study physician, Arthur Rosen, MD
* Hypertensive
* Taking medications (currently or within the last 3 months) known to influence appetite or metabolism
* Allergies to eggs
* Lactose intolerance
* Unwillingness to eat study foods
* Inability to travel to testing facility

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Increasing protein intake from lean beef/pork or soy/legumes sources will result in progressively decreased daily composite hunger and desire to eat, and increased fullness. The responses will not be different between groups of subjects. | 14 weeks

SECONDARY OUTCOMES:
Increasing the protein content of a test will result in progressively more robust and sustained changes in postprandial appetite and energy expenditure and blunted glycemic response. The responses will not be different between the groups of participants. | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Zhou J, Kim JE, Armstrong CL, Chen N, Campbell WW. Higher-protein diets improve indexes of sleep in energy-restricted overweight and obese adults: results from 2 randomized controlled trials. Am J Clin Nutr. 2016 Mar;103(3):766-74. doi: 10.3945/ajcn.115.124669. Epub 2016 Feb 10. PMID 26864362